CLINICAL TRIAL: NCT05043571
Title: Anti-CD7 Protein Expression Blocker (PEBL) Chimeric-Antigen Receptor (CAR) T-Cell Therapy for Relapsed/ Refractory T-Lineage Acute Lymphoblastic Leukaemia (CARTALL)
Brief Title: CARTALL: Chimeric-Antigen Receptor (CAR) T-Cell Therapy for Relapsed/ Refractory T-Lineage Acute Lymphoblastic Leukaemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/01325
Record Dates: First submitted 2021-06-13; First posted 2021-09-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-06

CONDITIONS: Lymphoblastic Leukemia, Acute, Childhood; Lymphoblastic Leukemia; Lymphoblastic Leukemia, Acute Adult; Lymphoblastic Leukemia in Children; CAR; CAR T-Cell-Related Encephalopathy Syndrome; Refractory Leukemia
Keywords: T-ALL; CAR-T cell therapy; CAR T-cell therapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Single arm Phase I Clinical Trial
  Interventions: Biological: CAR T-cell therapy

INTERVENTIONS:
Biological: CAR T-cell therapy — This is a single-centre, phase I study to determine the efficacy and safety of CAR T-cell therapy in patients with high-risk T-ALL, refractory or relapsed T-ALL.

SUMMARY:
The objective of this study is to assess the safety and efficacy of anti-CD7 CAR T-cells in patients with refractory or relapsed T-lineage acute lymphoblastic leukemia (T-ALL).

DETAILED DESCRIPTION:
A major obstacle to the development of effective CAR T-cells for T-cell malignancies is that the surface marker profile of malignant T-cells largely overlaps that of activated T lymphocytes. We developed a CAR T-cell approach that targets CD7, a T-cell marker highly expressed in all cases of T-cell ALL, including ETP-ALL. Its expression is also highly stable even in T-ALL cells exposed to chemotherapy. To prevent fratricide effect of the T cells, surface CD7 expression are effectively downregulated with the expression of an anti-CD7 Protein Expression Blocker (PEBL). Patients will receive anti-CD7 PEBL CART-cells. This will allow targeting the entire leukemia cell population to induce deeper and more durable remissions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis/ Disease define as:

  1. Relapsed T-cell acute lymphoblastic leukaemia/ lymphoma as defined by:

     Bone marrow disease = or > 0.01% by MRD as determined by flow cytometry

     Or CNS disease as defined as > 5 WBCs/ uL in CSF with morphological evidence of blasts or biopsy proven recurrence in the eye or brain

     Or Extramedullary relapse as defined by morphological evidence of blasts in the testis or any other extramedullary sites
  2. Induction failure as defined by:

     MRD = or > 1% by flow cytometry at the end of induction on day 33

     Or Failure to achieve morphological remission defined as > 5% blasts after standard induction chemotherapy
  3. Refractory disease as defined by:

     MRD = or > 0.01% by flow cytometry or molecular methods during 2 or more timepoints after induction therapy
* Minimum level of pulmonary reserve defined as Grade ≤ 1 dyspnoea and oxygen saturation (SpO2) of > 95% on room air
* Left ventricular systolic function (LVSF) ≥ 28% confirmed by echocardiogram, or left ventricular ejection fraction (LVEF) ≥ 45% confirmed by echocardiogram within 3 months of screening
* Karnofsky (age ≥ 16 years) or Lansky (age < 16 years) performance status ≥ 50 at screening
* Normal Age-adjusted eGFR Creatinine Clearance within 3 months of screening
* Alanine aminotransferase ≤ 5 times the upper limit of normal for age
* Patients with > 99% CD7 expression on blast cells will be eligible for anti-CD7 PEBL-CAR-T cell infusion.

Exclusion Criteria:

* Failure to meet any of the inclusion criteria
* Patients who test positive on urine pregnancy testing and are pregnant or are lactating
* Concomitant genetic syndromes associated with bone marrow failure states, such as Fanconi anaemia, Kostmann syndrome, Schwachman syndrome, or any other bone marrow failure syndrome with the exception of Down syndrome
* Prior malignancy, except carcinoma in situ of the skin or cervix treated with curative intent and no evidence of active disease
* Active or latent hepatitis B or hepatitis C infections within 8 weeks of screening, or any uncontrolled infection at screening
* Positive Human Immunodeficiency Virus (HIV) test within 8 weeks of screening
* Grade 2 to 4 acute graft-vs-host disease (GVHD) or extensive chronic GVHD
* Received an investigational medicinal product within 30 days of screening
* Central nervous system : Uncontrolled seizures or status epilepticus; increased intra-cranial pressure as evidenced by papilledema and CSF opening pressure > 20 cm water; decreased conscious state (any cause)

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-08 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participant who are flow cytometry minimal residual disease (MRD) negativity at 1 month after Anti-CD7 PEBL CAR T-cell infusion. | 30 days
  MRD levels will be determined by flow cytometry. The target sensitivity of flow MRD is <0.01% when available.

SECONDARY OUTCOMES:
Proportion of participant who are minimal residual disease (MRD) negative with molecular base assay at the end of 1 month after Anti-CD7 PEBL CAR T-cell infusion. | 30 days
  MRD levels will be determined by molecular based MRD by Ig/TCR. PCR and oncogene fusion transcript (OFT).
Proportion of patient who shows CAR T-cell persistence by immunophenotyping using flow cytometry in bone marrow, peripheral blood and CSF samples at multiple study time points following CAR T cell infusion | 1 month to 5 years
  Flow cytometry will be performed on bone marrow, peripheral blood and CSF samples at multiple study time points following CAR T cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Allen Yeoh, M.D, Principal Investigator — National University Hospital, Singapore; Dario Campana, M.D, PhD, Study Director — National University of Singapore
Locations (1):
- Allen Yeoh Eng Juh, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No